CLINICAL TRIAL: NCT03562104
Title: Swallowing Disorders and Consciousness Alteration in Severe Traumatic Brain Injury Patients
Brief Title: Swallowing Disorders in Minimally Consciousness Patients (MCS)
Acronym: TC-DEG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016/379 HP
Record Dates: First submitted 2018-05-25; First posted 2018-06-19 (Actual); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Swallowing Disorder; Traumatic Brain Injury
MeSH Terms: conditions — Deglutition Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Intervention Model Description: Description of swallowing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimally consciousness Patient (Experimental): Wessex Head Injury Matrix scale and Videofluoroscopy for characterization of swallowing disorders in Minimally consciousness Patient
  Interventions: Other: videofluoroscopy; Other: Wessex Head Injury Matrix scale

INTERVENTIONS:
Other: videofluoroscopy — Swallowing description in Minimally consciousness Patient
Other: Wessex Head Injury Matrix scale — Wessex Head Injury Matrix scale in Minimally consciousness Patient

SUMMARY:
This study aimed to characterize swallowing disorders in minimally consciousness patients after brain traumatic injury.

DETAILED DESCRIPTION:
After inclusion, the patients will underwent a videofluoroscopy and the Wessex Head Injury Matrix.

ELIGIBILITY:
Inclusion Criteria:

* Legal representant signed
* Aged between 18 and 70 years
* Having a severe TBI (Glasgow < 8)
* Without counterindication to underwent a VideoFluoroScopy
* Could hold a setting position

Exclusion Criteria:

* Pregnancy ongoing
* Having a pathologic al examination of IX, X, XII cranial nerve examination
* Massif faciale fracture
* Psychiatric illness
* Medical history of swallowing disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2019-06-01 (Estimated)

PRIMARY OUTCOMES:
Stages of swallowing disorders | Day 1
  swallowing disorder stage is done using videofluoroscopy

SECONDARY OUTCOMES:
Correlation between Wessex Head Injury Matrix (WHIM) and stage of swallowing disorder | Day 1
  Correlation between Wessex Head Injury Matrix (WHIM) and swallowing disorder (Videofluoroscopy)

CONTACTS AND LOCATIONS:
Overall Officials: Eric VERIN, Pr, Principal Investigator — University Hospital, Rouen
Locations (2):
- France (2):
  - Centre les Herbiers, Bois-Guillaume
  - UH Rouen, Rouen

IPD SHARING:
Plan to Share IPD: No